CLINICAL TRIAL: NCT04674020
Title: Registry for Migraine - Structural and Functional Magnetic Resonance Imaging Before and After Erenumab Treatment
Brief Title: Registry for Migraine - Structural and Functional MRI Before and After Erenumab Treatment
Acronym: REFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, Prinicipal Investigator, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-20033264
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-Arm (Experimental): Erenumab packed in a SureClick® Autoinjector Pen (AI).
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Erenumab 70 mg or 140 mg packed in a SureClick® Autoinjector Pen (AI)
  Other Names: Aimovig

SUMMARY:
This study aims to investigate structural and functional cerebral changes using magnetic resonance imaging before and after treatment with erenumab in patients with migraine.

DETAILED DESCRIPTION:
Migraine is a prevalent neurological disorder and a leading cause of years lived with disability worldwide. As of recent, therapies targeting calcitonin gene-related peptide (e.g. erenumab) have been approved for the preventive treatment of migraine. This study aims to investigate structural and functional cerebral changes using magnetic resonance imaging before and after treatment with erenumab in patients with migraine.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age greater than or equal to 18 years upon entry into screening
* History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self report
* Greater than or equal to 4 headache days that meet criteria as migraine days per month on average across the 3 months before screening after baseline period
* Must have demonstrated greater than or equal to 75% compliance in headache diary usage during baseline period

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

Disease Related

* Greater than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine headache
* Inability to differentiate between migraine from other headaches
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behaviour
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion Prior/Concomitant Therapy
* Previously received erenumab (Aimovig®)
* Received an anti-CGRP monoclonal antibody within 3 months prior to the start of the baseline period Prior/Concurrent Clinical Study Experience
* Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives since ending treatment on another investigational device or drug study (ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions

* Female subjects of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 16 weeks after the last dose of investigational product.
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 16 weeks after the last dose of investigational product.
* Evidence of current pregnancy or breastfeeding per subject self-report or medical records
* Subject has known sensitivity to any of the products or components to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge

Contraindications to MRI:

* Does not wish to be informed about unexpected MRI findings
* Severe claustrophobia
* Implanted magnetic material including pacemaker, prothesis, metal-clips, etc.
* Insulin pump which cannot be removed
* Magnetic foreign object in the body
* Surgical intervention within 6 weeks prior to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Headache Diary | Baseline Phase (Day -42 to -28) to Month 6]
  Headache diary with daily entries to record migraine-related data.

SECONDARY OUTCOMES:
3T Brain Structural and Functional Magnetic Resonance Imaging (MRI) at Baseline | Baseline Phase (Day -42 to -28)
  * MP2RAGE
  * GRAPPATINI
  * Gradient-Recalled-Echo (GRE) Sequence w/wo Magnetization Transfer (MT)
  * MPRAGE
  * Diffusion Tensor Imaging (DTI)
  * Resting State Functional MRI
  * Task-Based Functional MRI (visual stimulation with checkerboard)
  * 3D FLAIR
3T Brain Structural and Functional Magnetic Resonance Imaging (MRI) at Baseline at Month 6 | Week 24 ± 2 Weeks
  * MP2RAGE
  * GRAPPATINI
  * Gradient-Recalled-Echo (GRE) Sequence w/wo Magnetization Transfer (MT)
  * MPRAGE
  * Diffusion Tensor Imaging (DTI)
  * Resting State Functional MRI
  * Task-Based Functional MRI (visual stimulation with checkerboard)
  * 3D FLAIR
3T Brain Structural and Functional Magnetic Resonance Imaging (MRI) at Baseline at Month 12 | Week 48 ± 4 Weeks
  * MP2RAGE
  * GRAPPATINI
  * Gradient-Recalled-Echo (GRE) Sequence w/wo Magnetization Transfer (MT)
  * MPRAGE
  * Diffusion Tensor Imaging (DTI)
  * Resting State Functional MRI
  * Task-Based Functional MRI (visual stimulation with checkerboard)
  * 3D FLAIR
Headache Diary | Baseline Phase (Day -42 to -28) to Month 12
  Headache diary with daily entries to record migraine-related data.
Blood Specimen for Analysis of Biomarkers at Baseline | Baseline Phase (Day -42 to -28)
  * 31 mL Blood for Plasma
  * 16 mL Blood for Serum
  * 28 mL Blood for Heparinized Plasma
Blood Specimen for Analysis of Biomarkers at Month 6 | Week 24 ± 2 Weeks
  * 31 mL Blood for Plasma
  * 16 mL Blood for Serum
  * 28 mL Blood for Heparinized Plasma
Blood Specimen for Analysis of Biomarkers at Month 12 | Week 48 ± 4 Weeks
  * 31 mL Blood for Plasma
  * 16 mL Blood for Serum
  * 28 mL Blood for Heparinized Plasma
Semi-Structured Interview | Baseline Phase (Day -42 to -28)
  In-person semi-structured interview to record migraine-related data.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Denmark

REFERENCES:
- [Derived] Karlsson WK, Christensen RH, Al-Khazali HM, Kallemose T, Jawad BN, Andersen O, Ashina M, Ashina H. Plasma SuPAR and therapeutic response to erenumab in migraine: a REFORM study. J Headache Pain. 2025 Apr 24;26(1):86. doi: 10.1186/s10194-025-02037-9. PMID 40275185
- [Derived] Christensen RH, Ashina H, Al-Khazali HM, Zhang Y, Tolnai D, Poulsen AH, Cagol A, Hadjikhani N, Granziera C, Amin FM, Ashina M. Differences in Cortical Morphology in People With and Without Migraine: A Registry for Migraine (REFORM) MRI Study. Neurology. 2024 May;102(9):e209305. doi: 10.1212/WNL.0000000000209305. Epub 2024 Apr 17. PMID 38630960
- [Derived] Karlsson WK, Ashina H, Cullum CK, Christensen RH, Al-Khazali HM, Amin FM, Ashina M; REFORM Investigators. The Registry for Migraine (REFORM) study: methodology, demographics, and baseline clinical characteristics. J Headache Pain. 2023 Jun 12;24(1):70. doi: 10.1186/s10194-023-01604-2. PMID 37303034